CLINICAL TRIAL: NCT05094739
Title: Knowledge and Attitude of a Group of Egyptian Parents Toward Dental Treatment of Their Children During the Fourth Wave of COVID-19: A Cross Sectional Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Abd Elraheem Abd Elmonem Ismail, dentist, Cairo University
Other Study IDs: Covid 19
Record Dates: First submitted 2021-10-23; First posted 2021-10-26 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
title: Knowledge and Attitude of a group of Egyptian Parents toward Dental Treatment of their children during the Fourth Wave of COVID-19: A Cross Sectional Study.

aim: The aim of the study is to evaluate the knowledge and attitudes of a group of Egyptian parents toward dental treatment of their children during the fourth wave of COVID-19 pandemic.

DETAILED DESCRIPTION:
statement of the problem: COVID-19 is a global public health threat that affects the respiratory system and threatens millions of lives all over the world. The World Health Organization (WHO) declared on 30 Jan. 2020 that COVID-19 is a public health emergency (Clouthard et al. 2020).

Fear from infection transmission from person to person or from contaminated objects increased after emergence of COVID-19 as virus can survive in aerosols for 3 hours and on plastic and stainless steel surfaces up to 3 days (Surme et al. 2021).

As dentistry is a profession with high risk for transmission of COVID-19, it is affected greatly clinically and economically. Clinically as only cases which need immediate interference like trauma and swellings that obstruct the airway can be done, and routine dental care should be suspended. Economically this suspension of routine dental care causes closure of number of dental clinics due to real financial problems, anxiety and stress (Clouthard et al. 2020).

From patient's point of view, so many patients thought that dental clinics are dangerous areas as source of risk of infection with COVID-19 (Surme et al. 2021).

Rationale:

Coronavirus disease 2019 (COVID-19) is a great threat to global public health. More than 260 million confirmed cases have been reported according to the statistics of the World Health Organization (WHO), including over five million deaths. The original severe acute respiratory syndrome coronavirus that was identified at the end of 2019 had evolved and a variety of variants emerged. (WHO) has classified them into categories. Variants of concern include Alpha, Beta, Gamma and Delta. They all resulted in a new wave of pandemic and thousands of deaths. Lately a new variant named Omicron which immediately raised global concerns was considered as the fifth variant of concern by WHO On November 26, 2021(He et al. 2021).

So people must be aware about Corona virus and its variants to avoid the infection.COVID-19 is a long standing pandemic as the virus continuously mutates and new variants emerge which subsequently need new solutions.

Benefits:

1- Patient:

* Increasing awareness of patient and their parents toward COVID-19 and dentistry.

  2- Practitioner:
* Increasing the knowledge about the parents' attitude towards dental treatment during fourth wave of COVID-19 pandemic.

  3- Community:
* Increasing the knowledge and awareness of the community about COVID-19 pandemic (specially the fourth wave of COVID 19), and its relation with dentistry.

Aim of the study: is to evaluate the knowledge and attitudes of a group of Egyptian parents toward dental treatment of their children during the fourth wave of COVID-19 pandemic.

PO format:

* P: A group of Egyptian parents.
* O: Knowledge and attitude of a group of Egyptian parents toward dental treatment of their children during the fourth wave of COVID-19 pandemic.

Primary outcome: Knowledge and attitude of a group of Egyptian parents toward dental treatment of their children during the fourth wave of COVID-19 pandemic.

Measurement method: Questionnaire by (Deema& Nada Farsi, 2021), Developed from ( Yip et al. 2007)& (Sun et al. 2020)

Unit of measurement:

* Binary question (Yes, No)
* Close-ended questions.

Secondary outcome:

1. Attitudes regarding taking children to see a dentist during the fourth wave of COVID-19 pandemic.

   Measurement method: Questionnaire by (Deema& Nada Farsi, 2021) Developed from ( Yip et al. 2007)& (Sun et al. 2020)

   Unit of measurement:

   -Binary question (Yes, No)

   - Close-ended questions.
2. Attitudes regarding maintenance of next visits during fourth wave of COVID-19 pandemic.

   Measurement method: Direct question

   Unit of measurement:

   -Binary question (Yes, No)

   Methods:

   A) Study design and setting.
   * Study design Cross-sectional study
   * Settings:

     _ Location: Clinics of Paediatric dentistry and Dental Public Health Department, Faculty of dentistry, Cairo University.

     _ Methodology:

     • The questionnaires will be distributed and filled under supervision of the primary investigator.

     • Each parent will be allowed to fulfill the questionnaire.

     • The parents will answer the questions in the questionnaire (Arabic version).

     • The questionnaire was developed from (Yip et al. 2007) & (Sun et al. 2020).

     • The questionnaire was then modified and validated by (Deema& Nada Farsi, 2021).

     • Then the author chose some of the questions of the questionnaire (with a reduced number) to be matched with the concept of the study.

     • All the questionnaires are translated into Arabic language

   B) Participants
   * Eligibility criteria and selection methods:

   Inclusion criteria:

   -Parents with at least intermediate education.

   Exclusion criteria:
   * Illiterate parents.
   * Refusal of participation

   C) Variables:
   * Details about variables:

   Primary outcome: Knowledge and attitude of a group of Egyptian parents toward dental treatment of their children during the fourth wave of COVID-19 pandemic.

   Measurement method: Questionnaire by (Deema& Nada Farsi, 2021), Developed from ( Yip et al. 2007)& (Sun et al. 2020)

   Unit of measurement:

   -Binary question (Yes, No)

   - Close-ended questions.

   Secondary outcome:1- Attitudes regarding taking children to see a dentist during the fourth wave of COVID-19 pandemic.

   Measurement method: Questionnaire by (Deema& Nada Farsi, 2021) Developed from ( Yip et al. 2007)& (Sun et al. 2020)

   Unit of measurement:

   -Binary question (Yes, No)

   - Close-ended questions.

2- Attitudes regarding maintenance of next visits during fourth wave of COVID-19 pandemic.

Measurement method: Direct question

Unit of measurement:

-Binary question (Yes, No).

_Potential confounders: Age, sex, degree of awareness, degree of education, parental dental anxiety due to COVID-19 Pandemic.

_Data sources and management:

Data will be obtained through written questionnaires for assessing Knowledge and Attitude of a group of Egyptian Parents toward Dental Treatment of their children during the Fourth Wave of COVID-19. Data collected will be saved and tabulated on computer for back up and finally statistically analysed.

_ Addressing potential sources of bias:

Selection bias:

All parents fulfilling the inclusion criteria, attending the days of examination will be included.

Information bias:

Information bias will be avoided by explaining to the parents the aim of the study without guiding them to specific answers.

Reporting bias:

All outcomes will be reported.

D) Study size:

- Study size:

A power analysis was designed to have adequate power to apply a statistical test of the research question regarding the knowledge and attitude of a group of Egyptian parents toward dental treatment of their children during the fourth wave of COVID-19 pandemic. According to the results of a previous study -in which the prevalence of good knowledge was (42.4%)- and by adopting a confidence interval of (95%), a margin of error of (5%) with finite population correction; The predicted sample size (n) was a total of (375) cases. Sample size calculation was performed using Epi info for windows version 7.2 .

E) Quantitative variables :

-Handling of quantitative variables in the analysis Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data was found to be normally distributed, it will be presented as mean and standard deviation values. If the assumption of normality was found to be violated, the data will be presented as median and range values.

Handling of categorical/ qualitative variables:

Categorical data will be represented as frequency (n) and percentage (%).

F) Statistical methods:

- Statistical methods: Categorical data will be represented as frequency (n) and percentage (%) and will be analyzed using chi square test. Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data was found to be normally distributed, it will be presented as mean and standard deviation values and independent t-test will be used for the analysis. If the assumption of normality was found to be violated; the data will be presented as median and range values and will be analyzed using Mann-Whitney U test. The significance level will be set at P ≤0.05 for all tests. Statistical analysis will be performed with IBM SPSS Statistics Version 26 for Windows.

References:

1. Farsi, D., & Farsi, N. (2021). Mothers' Knowledge, Attitudes, and Fears About Dental Visits During the COVID-19 Pandemic: A Cross-sectional Study. Journal of International Society of Preventive & Community Dentistry, 11(1), 83.
2. Surme, K., Akman, H., Akbaydogan, L. C., & Akin, M. (2021). Evaluation of Parents' Knowledge and Attitudes Towards Pediatric Dental Practice during the COVID-19 Pandemic. Oral Health & Preventive Dentistry, 19(1), 271-277.
3. Sun, J., Xu, Y., Qu, Q., & Luo, W. (2020). Knowledge of and attitudes toward COVID-19 among parents of child dental patients during the outbreak. Brazilian oral research, 34.
4. Yip HK, Tsang PC, Samaranayake LP, Li AH. Knowledge of and attitudes toward severe acute respiratory syndrome among a cohort of dental patients in Hong Kong following a major local outbreak. Community Dent Health. 2007;24:43-8.
5. Barghout, N., Al Habashneh, R., Ryalat, S. T., Asa'ad, F. A., & Marashdeh, M. (2012). Patients' perception of cross-infection prevention in dentistry in Jordan. Oral Health and Preventive Dentistry, 10(1), 9.
6. World Health Organization. (2020). Coronavirus disease (COVID-19): How is it transmitted. Geneva, Switzerland: WHO.

   ( https://www.who.int/emergencies/diseases/novel-coronavirus-2019/question-and-answers-hub/q-a-detail/coronavirus-disease-covid-19-how-is-it-transmitted)
7. World Health Organization. (2020). Coronavirus disease ( COVID-19). ( https://www.who.int/emergencies/diseases/novel-coronavirus-2019/question-and-answers-hub/q-a-detail/coronavirus-disease-covid-19)
8. Coulthard, P., Thomson, P., Dave, M., Coulthard, F. P., Seoudi, N., & Hill, M. (2020). The COVID-19 pandemic and dentistry: the clinical, legal and economic consequences-part 1: clinical. British Dental Journal, 229(11), 743-747.
9. Coulthard, P., Thomson, P., Dave, M., Coulthard, F. P., Seoudi, N., & Hill, M. (2020). The COVID-19 pandemic and dentistry: the clinical, legal and economic consequences-part 2: consequences of withholding dental care. British Dental Journal, 229(12), 801-805.
10. He, X., Hong, W., Pan, X., Lu, G., & Wei, X. (2021). SARS-CoV-2 Omicron variant: characteristics and prevention. MedComm.

    (https://onlinelibrary.wiley.com/doi/full/10.1002/mco2.110)
11. Parvaie, P., & Osmani, F. (2022). Dentistry during COVID-19: patients' knowledge and satisfaction toward health protocols COVID-19 during dental treatment. European journal of medical research, 27(1), 1-7.

ELIGIBILITY:
Inclusion Criteria:

* Parents with at least intermediate educational level.

Exclusion Criteria:

* Illiterate parents.
* Refusal of participation

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: -Parents with at least an intermediate educational level and aware about COVID-19 and their attitudes toward dental treatments of their children
Sampling Method: Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Knowledge and attitude of a group of Egyptian parents toward dental treatment of their children during the fourth wave of COVID-19 pandemic. | 12 months
  * Binary question (Yes, No).
  * close-ended questions

SECONDARY OUTCOMES:
1-Attitudes regarding taking children to see a dentist during the fourth wave of COVID-19 pandemic. 2-Attitudes regarding maintenance of next visits during fourth wave of COVID-19 pandemic | 12 months
  * Binary question (Yes, No).
  * close-ended questions

REFERENCES:
- See also: Mothers' Knowledge, Attitudes, and Fears About Dental Visits During the COVID-19 Pandemic: A Cross-sectional Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7934827/
- See also: Evaluation of Parents' Knowledge and Attitudes Towards Pediatric Dental Practice during the COVID-19 Pandemic — http://www.quintpub.com/journals/ohpd/fulltext.php?article_id=21403